CLINICAL TRIAL: NCT05708144
Title: Study of a Novel Near-infrared(NIR) Fluorescent Molecular Probe Targeting Trop-2 for the Identification of Benign and Malignant Breast Tissue
Brief Title: NIR Fluorescent Molecular Probe for the Identification of Breast Tissue
Acronym: NIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiang'an Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Weiling Chen，MD, attending doctor, Xiang'an Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XianganHXiamenU
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: breast tissue; NIR-II; Trop-2; diagnosis
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indocyanine green-Sacituzumab govitecan-hziy (ICG-SG) (Experimental): The fresh excision breast cancer tissues were completely soaked in the ICG-SG incubation solution for about 10 minutes, followed by 5 minutes of rinsing with PBS buffer and drying with the use of absorbent paper. Then fluorescence imaging was performed with the DPM NIR-II system. And the result was analyzed to identify the tumor area and distinguish the tumor boundary.
  Interventions: Diagnostic Test: ICG-SG incubation solution

INTERVENTIONS:
Diagnostic Test: ICG-SG incubation solution — The fresh excision breast cancer tissues were completely soaked in the incubation solution and performed fluorescence imaging.

SUMMARY:
Accurate evaluation of tumor boundaries in breast-conserving surgery is critical to reducing the second operation of patients. Near-infrared (NIR) fluorescence imaging using molecular agents has shown promise for in situ imaging during resection. However, very effective probes can be applied to clinical trials up to now, which limits the clinical application of fluorescence imaging. Here we developed a new technology that can quickly identify the tumor area of the resected breast tissue during the operation and distinguish the tumor boundary. In brief, the breast tissues were incubated with the probe immediately after intraoperative resection and imaged to identify the tumor area and distinguish the tumor boundary. The accuracy of fluorescence imaging was confirmed by pathological diagnosis.

DETAILED DESCRIPTION:
After enrollment, the patients received surgical treatment according to clinical diagnosis and treatment. During the operation, the excised breast tissue was incubated, and the specific procedure was as follows.

1. Preparation of the incubation solution: The probe was dissolved in phosphate buffer saline(PBS) buffer as the incubation solution at room temperature in the dark.
2. In vitro incubation of fresh breast cancer tissues: The fresh excision breast cancer tissues were completely soaked in the incubation solution for about 10 minutes, followed by 5 minutes rinse with PBS buffer and drying with the use of absorbent paper.
3. Analysis of the images in the "Digital Precision Medicine(DPM)" NIR-II system. The DPM parameter was set up before scaling. Then fluorescence imaging was performed with the DPM NIR-II system. And the result was analyzed to identify the tumor area and distinguish the tumor boundary.
4. Confirmed the diagnosis by pathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age; Female; Patients presenting with a breast nodule or mass presumed to be resectable on pre-operative assessment; Good operative candidate; Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

* Patients unable to participate in the consent process; Patients had contraindications to surgery, such as serious cardiopulmonary disease, coagulation dysfunction, etc; Other conditions that the researcher considers inappropriate to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Expression of the trop-2 in the tumor | 2 years
  Ability of the imaging system to detect the expression of the trop-2 in the mass (i.e tumor).
Uptake of the dye by the tumor | 2 years
  Ability of the imaging system to discern the uptake of the dye by the tumor. Detected with imaging probe.
False positive rates of ICG-SG | 2 years
  Microscopic examination and immunohistochemistry of tumor performed by a pathologist. This will allow investigators to compare pathology results with fluorescence images taken by imaging probe to calculate false positive (i.e., identification of non Trop2-positive tumors) rates of ICG-SG.

SECONDARY OUTCOMES:
Incidence rates of all adverse events (AEs) | 2 years
  Tissue incubation adverse events and adverse device events (ADEs)

CONTACTS AND LOCATIONS:
Overall Officials: Guojun Zhang, MD, Study Director — Xiang'an Hospital of Xiamen University
Locations (1):
- Xiamen Key Laboratory of Endocrine-Related Cancer Precision Medicine, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li C, Mi J, Wang Y, Zhang Z, Guo X, Zhou J, Hu Z, Tian J. New and effective EGFR-targeted fluorescence imaging technology for intraoperative rapid determination of lung cancer in freshly isolated tissue. Eur J Nucl Med Mol Imaging. 2023 Jan;50(2):494-507. doi: 10.1007/s00259-022-05975-7. Epub 2022 Oct 8. PMID 36207638
- See also: A new fluorescence imaging technology for intraoperative rapid determination of lung cancer in freshly isolated tissue — http://pubmed.ncbi.nlm.nih.gov/36207638/